CLINICAL TRIAL: NCT00479232
Title: A Phase I Clinical Trial of Vorinostat in Combination With Decitabine in Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Phase I Trial of Vorinostat (MK-0683, SAHA) in Combination With Decitabine in Patients With AML or MDS (MK-0683-055 EXT1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-055; 2007_500
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2011-08-31 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Leukemia, Myelocytic, Acute Myelodysplastic Syndromes; Myelodysplastic Syndromes
Keywords: Leukemia; Myelocytic; Acute Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Vorinostat; Decitabine

ARMS (2):
- Cohort 1: Vorinostat (sequential) (Experimental): Vorinostat 400 mg capsules once daily given 7, 10 or 14 days in 28 day cycles. Up to 24 months of treatment.
  Decitabine IV 20 mg/m^2 daily for 5 days in each 28 day cycle. Up to 24 months of treatment.
  Interventions: Drug: vorinostat; Drug: decitabine
- Cohort 2: Vorinostat (concurrent) (Experimental): Vorinostat 400 mg capsules once daily given 7 days, 14 days with 8 day break after first 7 days or 14 days without break, out of 28 day cycles.
  Decitabine IV 20 mg/m^2 daily for 5 days in each 28 day cycle. Up to 24 months of treatment.
  Interventions: Drug: vorinostat; Drug: decitabine

INTERVENTIONS:
Drug: vorinostat
  Other Names: MK-0683; SAHA
Drug: decitabine
  Other Names: Dacogen

SUMMARY:
This study is to evaluate the safety and tolerability of vorinostat in combination with decitabine as well as the in vivo molecular and biological effects of vorinostat in patients with refractory or relapsed Acute Myelogenous Leukemia (AML) and intermediate or high risk as defined by International Prognostic Scoring System (IPSS) Myelodysplastic Syndrome (MDS). Participants with Acute Myelogenous Leukemia or Myelodysplastic Syndrome are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old with refractory/relapsed AML

  * If untreated AML, patient is older than 60 years old and not a candidate for standard chemotherapy
* Patient is at least 4 weeks from prior treatment and has recovered from all prior treatment side effects
* Patient has no known liver or kidney problems
* Patient knows of no reason they can not receive transfusions of blood clotting cells (platelets)
* Patient is able to swallow capsules
* Patients both male and female are willing to practice birth control during the study

Exclusion Criteria:

* Patient has received prior treatment with valproic acid, decitabine or azacitidine
* Being is less than 18 years of age or if patient has untreated AML is below 60 years of age
* Patient is a women who is pregnant or breastfeeding. Patient has an active infection that requires antibiotics
* Patient has uncontrolled illness including but not limited to the following: heart problems (congestive heart failure, unstable angina pectoris, cardiac arrhythmia), inflammation of the pancreas; a mental or social condition that may interfere with patient following study procedures
* Patient has known human immunodeficiency virus (HIV) infection or HIV-related malignancy. Patient has a known history of hepatitis B or C infection
* Patient currently has another active cancer other than certain types of skin cancer
* Patient is heterosexual and able to have a child and is unwilling to practice birth control during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kirschbaum M, Gojo I, Goldberg SL, Bredeson C, Kujawski LA, Yang A, Marks P, Frankel P, Sun X, Tosolini A, Eid JE, Lubiniecki GM, Issa JP. A phase 1 clinical trial of vorinostat in combination with decitabine in patients with acute myeloid leukaemia or myelodysplastic syndrome. Br J Haematol. 2014 Oct;167(2):185-93. doi: 10.1111/bjh.13016. Epub 2014 Jul 8. PMID 25040094

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent, Vorinostat 400mg qd x 7d/4wk + Decitabine: (concurrent) vorinostat 400 mg capsules given once daily (qd) on Days 1 to 7 in a 28 day cycle, along with decitabine intravenous (IV) 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400mg qd x 7d/2wk + Decitabine: (concurrent) vorinostat 400 mg capsules given qd on Days 1 to 7 and Days 15 to 21 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD): (concurrent) vorinostat 400 mg capsules given qd on Days 1 to 14 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 7d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given qd on Days 6 to 12 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 10d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given qd on Days 6 to 15 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD): (sequential) vorinostat 400 mg capsules given qd on Days 6 to 19 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
Period: Overall Study
Arm/Group | Concurrent, Vorinostat 400mg qd x 7d/4wk + Decitabine | Concurrent, Vorinostat 400mg qd x 7d/2wk + Decitabine | Concurrent, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD) | Sequential, Vorinostat 400mg qd x 7d/4wk + Decitabine | Sequential, Vorinostat 400mg qd x 10d/4wk + Decitabine | Sequential, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD)
Started | 3 | 3 | 28 | 3 | 4 | 30
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 28 | 3 | 4 | 30
Not completed — Adverse Event | 0 | 0 | 5 | 0 | 0 | 10
Not completed — Deviation from Protocol | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Progressive Disease | 3 | 1 | 12 | 3 | 3 | 12
Not completed — Withdrew Consent | 0 | 2 | 6 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat + Decitabine, Concurrent: (concurrent) Vorinostat 400 mg capsules once daily given 7 days, 14 days with 8 day break after first 7 days or 14 days without break, out of 28 day cycles along with decitabine IV 20 mg/m^2 daily for 5 days in each 28 day cycle. Up to 24 months of treatment.
- Vorinostat + Decitabine, Sequential: (sequential) Vorinostat 400 mg capsules once daily given 7, 10 or 14 days in 28 day cycles along with decitabine IV 20 mg/m^2 daily for 5 days in each 28 day cycle. Up to 24 months of treatment.
- Total: Total of all reporting groups
Arm/Group | Vorinostat + Decitabine, Concurrent | Vorinostat + Decitabine, Sequential | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (13.0) | 66.6 (13.8) | 65.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity (DLT) Events
Description: Participants who received at least one dose of vorinostat in combination with decitabine intravenous (IV) at a dose of 20 mg/m^2 daily for 5 days along with oral vorinostat 400 mg once daily for 7 to 14 days in a 28-day cycle concurrently or sequentially, were evaluated to determine the maximum tolerable dose (MTD) determined by the number of participants experiencing dose limiting toxicity (DLT) events defined as any Grade 3 or 4 non-hematological toxicity (reported adverse event) and/or myelosuppression lasting >42 days.
Time Frame: Day 1 to 28 of Cycle 1
Measure: Number; unit: participants
Groups:
- Concurrent, Vorinostat 400mg qd x 7d/4wk + Decitabine: (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 7 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400mg qd x 7d/2wk + Decitabine: (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 7 and Days 15 to 21 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD): (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 14 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 7d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given once daily on Days 6 to 12 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 10d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given once daily on Days 6 to 15 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD): (sequential) vorinostat 400 mg capsules given once daily on Days 6 to 19 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
Arm/Group | Concurrent, Vorinostat 400mg qd x 7d/4wk + Decitabine | Concurrent, Vorinostat 400mg qd x 7d/2wk + Decitabine | Concurrent, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD) | Sequential, Vorinostat 400mg qd x 7d/4wk + Decitabine | Sequential, Vorinostat 400mg qd x 10d/4wk + Decitabine | Sequential, Vorinostat 400mg qd x 14d/4wk + Decitabine (MTD)
Number analyzed (Participants) | 3 | 3 | 28 | 3 | 4 | 30
participants | 0 | 0 | 0 | 0 | 0 | 1

2. Other Pre Specified Outcome: Objective Response Rate in Participants Treated With Vorinostat + Decitabine With Refractory or Relapse Acute Myelogenous Leukemia (AML)
Description: Objective Response Rate was measured in participants with refractory or relapse AML (acute myelogenous leukemia) in combination with Decitabine who were treated with vorinostat and decitabine on either a concurrent or sequential regimen. The Objective response was defined as any confirmed complete remission or any confirmed partial remission for AML participants and complete remission, confirmed partial remission or confirmed hematologic improvement for Myelodysplastic Syndrome (MDS) participants.
Time Frame: Approximately 6 months
Measure: Number; unit: percentage of participants
Groups:
- Refractory or Relapsed AML, Concurrent: Participants with Refractory or Relapsed AML who were treated with vorinostat and Decitabine concurrently.
- Refractory or Relapsed AML, Sequential: Participants with Refractory or Relapsed AML who were treated with vorinostat and Decitabine sequentially.
Arm/Group | Refractory or Relapsed AML, Concurrent | Refractory or Relapsed AML, Sequential
Number analyzed (Participants) | 14 | 15
percentage of participants | 7.1 (0) [0.2 to 33.9] | 0.0 (NA) [0.0 to 21.8]

3. Other Pre Specified Outcome: Objective Response Rate in Participants Treated With Vorinostat + Decitabine With Intermediate-high Risk Myelodysplastic Syndrome (MDS) or Untreated Acute Myelogenous Leukemia (AML)
Description: Objective Response Rate was measured in participants with intermediate-high risk MDS or untreated AML who were treated with vorinostat and decitabine either on a concurrent or sequential regimen. The Objective response was defined as any confirmed complete remission or any confirmed partial remission for AML participants and complete remission, confirmed partial remission or confirmed hematologic improvement for MDS participants.
Time Frame: Approximately 6 months
Measure: Number; unit: percentage of participants
Groups:
- Untreated AML or Intermediate, Concurrent: Participants with Untreated AML or Intermediate-High
  Risk MDS who were treated with vorinostat and Decitabine
  concurrently.
- Untreated AML or Intermediate, Sequential: Participants with Untreated AML or Intermediate-High
  Risk MDS who were treated with vorinostat and Decitabine
  sequentially.
Arm/Group | Untreated AML or Intermediate, Concurrent | Untreated AML or Intermediate, Sequential
Number analyzed (Participants) | 20 | 22
percentage of participants | 35.0 (170.3) | 13.6 (119.2)

ADVERSE EVENTS:
Groups:
- Concurrent, Vorinostat 400 mg qd x 7d/4wk + Decitabine: (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 7 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400 mg qd x 7d/2wk + Decitabine: (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 7 and Days 15 to 21 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Concurrent, Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD): (concurrent) vorinostat 400 mg capsules given once daily on Days 1 to 14 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400 mg qd x 7d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given once daily on Days 6 to 12 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential, Vorinostat 400 mg qd x 10d/4wk + Decitabine: (sequential) vorinostat 400 mg capsules given once daily on Days 6 to 15 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
- Sequential,Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD): (sequential) orinostat 400 mg capsules given once daily on Days 6 to 19 in a 28 day cycle, along with decitabine IV 20mg/m^2 daily for 5 days in each 28 day cycle, up to 24 months of treatment.
Arm/Group | Concurrent, Vorinostat 400 mg qd x 7d/4wk + Decitabine | Concurrent, Vorinostat 400 mg qd x 7d/2wk + Decitabine | Concurrent, Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD) | Sequential, Vorinostat 400 mg qd x 7d/4wk + Decitabine | Sequential, Vorinostat 400 mg qd x 10d/4wk + Decitabine | Sequential,Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD)
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 21/28 | 2/3 | 4/4 | 25/31
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 27/28 | 3/3 | 4/4 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent, Vorinostat 400 mg qd x 7d/4wk + Decitabine (N=3) | Concurrent, Vorinostat 400 mg qd x 7d/2wk + Decitabine (N=3) | Concurrent, Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD) (N=28) | Sequential, Vorinostat 400 mg qd x 7d/4wk + Decitabine (N=3) | Sequential, Vorinostat 400 mg qd x 10d/4wk + Decitabine (N=4) | Sequential,Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 12 (16) | 1 (1) | 1 (1) | 7 (8)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (5)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 6 (7) | 0 (0) | 2 (4) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent, Vorinostat 400 mg qd x 7d/4wk + Decitabine (N=3) | Concurrent, Vorinostat 400 mg qd x 7d/2wk + Decitabine (N=3) | Concurrent, Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD) (N=28) | Sequential, Vorinostat 400 mg qd x 7d/4wk + Decitabine (N=3) | Sequential, Vorinostat 400 mg qd x 10d/4wk + Decitabine (N=4) | Sequential,Vorinostat 400 mg qd x 14d/4wk + Decitabine (MTD) (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (3) | 3 (6) | 2 (2) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (4)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (10) | 8 (17) | 2 (4) | 1 (1) | 3 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 9 (20) | 0 (0) | 0 (0) | 6 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 11 (31) | 1 (2) | 1 (1) | 8 (20)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (7) | 1 (1) | 1 (3) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 16 (24) | 1 (2) | 3 (5) | 11 (15)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 16 (25) | 1 (1) | 3 (3) | 15 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 3 (3)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (2) | 17 (29) | 3 (3) | 3 (4) | 20 (25)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 10 (15) | 2 (2) | 2 (3) | 11 (12)
Asthenia (General disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 2 (2) | 4 (4)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 11 (12) | 1 (1) | 1 (2) | 2 (3)
Fatigue (General disorders) | 3 (3) | 1 (1) | 11 (20) | 2 (2) | 3 (4) | 19 (24)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 7 (9)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 7 (9) | 0 (0) | 0 (0) | 5 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 7 (10) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 2 (17)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (7)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (3)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 2 (4)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Granulocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 9 (14) | 2 (2) | 1 (1) | 10 (13)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemosiderosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6) | 2 (4) | 1 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 5 (6) | 2 (2) | 1 (1) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 2 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (13) | 2 (2) | 1 (1) | 6 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (8) | 2 (2) | 1 (1) | 4 (5)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (5) | 3 (4) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 3 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 4 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 11 (16) | 0 (0) | 1 (1) | 7 (9)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (3) | 7 (9) | 1 (1) | 0 (0) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Testis discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 6 (6) | 1 (1) | 2 (2) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 6 (6)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 2 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 4 (4)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 4 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.